CLINICAL TRIAL: NCT03493308
Title: Pain Neuroscience Education and Exercise in Institutionalized Older Adults With Pain: A Feasibility Study
Brief Title: Pain Neuroscience Education and Exercise in Institutionalized Older Adults With Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Assistant Professor, Aveiro University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 09-CED/2018
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain neuroscience and exercise (Experimental): Participants will received an 8 week intervention consisting of pain neuroscience education and exercise. Pain neuroscience education will be conducted in line with international guidelines, covering the neurophysiology of pain, transition from from acute to chronic pain and the nervous system ability to modulate the pain experience. exercise will include general exercise and dance.
  Interventions: Other: Pain neuroscience education; Other: Exercise

INTERVENTIONS:
Other: Pain neuroscience education — PNE will be conducted in line with international guidelines and will cover the neurophysiology of pain, transition from acute to chronic pain and the nervous system ability to modulate the pain experience.
Other: Exercise — Exercise will be provided in different formats including general exercise, strengthening, dance.

SUMMARY:
The primary objectives of this study are to:

* Evaluate recruitment procedures and adherence rates;
* Evaluate the ability to understand the concepts of pain neurophysiology;
* Evaluate the acceptability of an intervention program based on pain neuroscience education and exercise by institutionalized older adults and the institutions where they are.

DETAILED DESCRIPTION:
Participants will be older adults with pain that are institutionalized and assess the feasibility of implementing an intervention consisting of pain neuroscience education in addition to exercise. It is antecipated that the intervention will consist of 1 to 2 sessions per week during 8 weeks and will be delivered in small groups. Participants will be assessed for pain intensity, duration, catastrophizing, fear of movement, knowledge of pain neuroscience, depression and performance.

ELIGIBILITY:
Inclusion Criteria:

* Be institutionalized in any type of response (nursing home, day care, ...), be able to read and write, have chronic pain (defined as pain lasting 3 months or more and felt at least once a week during these 3 months ) anywhere in the body, and have a statement from the institution's physician authorizing participation in the exercise sessions.

Exclusion Criteria:

* Have any contra-indication to exercise and have cognitive limitations (evaluated through the Montreal Cognitive Assessment questionnaire).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Assessed using the vertical numeric rating scale that assesses pain intensity (range 0-10 and higher values are indicative of higher pain intensity)
Pain intensity | 9 weeks
  Assessed using the vertical numeric rating scale that assesses pain intensity (range 0-10 and higher values are indicative of higher pain intensity)
Pain intensity | 3 months
  Assessed using the vertical numeric rating scale that assesses pain intensity (range 0-10 and higher values are indicative of higher pain intensity)

SECONDARY OUTCOMES:
Pain location | Baseline
  Assessed using a body chart where the patients identifies the painful body segments
Pain location | 9 weeks
  Assessed using a body chart where the patients identifies the painful body segments
Pain location | 3 months
  Assessed using a body chart where the patients identifies the painful body segments
Pain frequency | Baseline
  Assessed using a closed question on pain frequency for the last week
Pain frequency | 9 weeks
  Assessed using a closed question on pain frequency for the last week
Pain frequency | 3 months
  Assessed using a closed question on pain frequency for the last week
Depression | Baseline
  Assessed using the Geriatric Depression Scale (range 0-15 and values of 5 or higher are indicative of depression)
Depression | 9 weeks
  Assessed using the Geriatric Depression Scale (range 0-15 and values of 5 or higher are indicative of depression)
Depression | 3 months
  Assessed using the Geriatric Depression Scale (range 0-15 and values of 5 or higher are indicative of depression)
Knowledge of pain neuroscience | Baseline
  Assessed using the pain neurophysiology questionnaire
Knowledge of pain neuroscience | 9 weeks
  Assessed using the pain neurophysiology questionnaire (range 0-19 and higher values are indicative of more knowledge on pain neurophysiology)
Knowledge of pain neuroscience | 3 months
  Assessed using the pain neurophysiology questionnaire (range 0-19 and higher values are indicative of more knowledge on pain neurophysiology)
Pain catastrophizing | Baseline
  assessed using the Pain Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Pain catastrophizing | 9 weeks
  assessed using the Pain Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Pain catastrophizing | 3 months
  assessed using the Pain Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Fear of movement | Baseline
  Assessed using the TAMPA Scale, which assesses fear of movement (range: 13-52 and higher values are indicative of higher levels of fear of movement)
Fear of movement | 9 weeks
  Assessed using the TAMPA Scale (range: 13-52 and higher values are indicative of higher levels of fear of movement)
Fear of movement | 3 months
  Assessed using the TAMPA Scale (range: 13-52 and higher values are indicative of higher levels of fear of movement)
Gait velocity | Baseline
  Assessed using the gait velocity test - the time, in seconds, that each participant takes to walk 4 meters
Gait velocity | 9 weeks
  Assessed using the gait velocity test - the time, in seconds, that each participant takes to walk 4 meters
Gait velocity | 3 months
  Assessed using the gait velocity test - the time, in seconds, that each participant takes to walk 4 meters
Postural control | Baseline
  Assessed using the Timed up and go test - the time, in seconds, that it takes to stand from a chair, walk 3 meters, turn, walk another 3 meters to sit in the chair.
Postural control | 9 weeks
  Assessed using the Timed up and go test - the time, in seconds, that it takes to stand from a chair, walk 3 meters, turn, walk another 3 meters to sit in the chair.
Postural control | 3 months
  Assessed using the Timed up and go test - the time, in seconds, that it takes to stand from a chair, walk 3 meters, turn, walk another 3 meters to sit in the chair.

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Silva, PhD, Principal Investigator — Aveiro University
Locations (1):
- Lar de Fermentelos, Águeda Municipality, Portugal

IPD SHARING:
Plan to Share IPD: No